CLINICAL TRIAL: NCT01668290
Title: Assessment of Patients With Suspected CAD: What is the Best Initial Imaging Strategy? Cardiac Computed Tomographic Angiography,(CCTA) vs Stress Echocardiography (SE) vs SPECT
Brief Title: Assessment of Patients With Suspected Coronary Artery Disease (CAD): What is the Best Initial Imaging Strategy?
Acronym: IMAGE-CAD
Status: Completed | Type: Observational
Sponsor: Harald Becher (Other)
Collaborators: Alberta Health services (Other); University of Alberta (Other)
Responsible Party: Sponsor-Investigator, Harald Becher, Heart and Stroke Foundation Chair for Cardiovascular Research, University of Alberta
Organization: University of Alberta (Other)
Other Study IDs: CMI 1D; Pro00026591 (Other: Health Research Ethics Board)
Record Dates: First submitted 2012-08-13; First posted 2012-08-20 (Estimated); Last update posted 2017-03-16 (Actual); Status verified 2017-03

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Stress Echocardiography; Single Photon Emission Computed Tomography; Cardiac Computed Tomographic Angiography; outcomes
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Stress Echocardiography: Patients will be randomized to one of three imaging modalities. One imaging modality thay can be randomized to is Stress Echocardiography.
- SPECT: Patients will be randomized to one of three imaging modalities. One imaging modality thay can be randomized to is Single Photon Emission Computed Tomography (SPECT)
- CCTA: Patients will be randomized to one of three imaging modalities. One imaging modality thay can be randomized to is Cardiac Computed Tomographic Angiography (CCTA)

SUMMARY:
Patients who present with chest pain are investigated with tests designed to confirm or exclude the presence of Coronary Artery Disease (CAD), as well as determine risk of poor outcome. It is not known which imaging test would be best when used first for investigating a patient presenting with exertional chest pain. This trial is designed to compare outcomes of the use of coronary CT, stress echocardiography and nuclear perfusion (SPECT) in a pilot study. Patients with no history of coronary disease presenting with chest pain will be randomly assigned to one of the three test modalities as the initial imaging test. The three imaging strategies will be compared regarding the subsequent use of healthcare resources over a year.

DETAILED DESCRIPTION:
This is a pilot study on imaging strategies for diagnosis of coronary artery disease. The pilot trial aims to answer the question "Which non-invasive test (single photon emission computed tomography (SPECT), stress echocardiography or coronary CT angiography (CCTA)) is the best first test in suspected coronary artery disease with respect to patient outcome and downstream health costs?" Patients are randomly assigned to one of the imaging modalities. All imaging and therapeutic procedures in this trial are clinically indicated. The only change from standard patient management is the selection of the initial imaging test. Instead of leaving the selection of the initial imaging test to the referring physician (whose decision is not evidence based), patients presenting with chest pain that fall into the inclusion/exclusion criteria of the study will be randomly assigned to one of the imaging modalities. Patients will also be followed at 1, 6 and 12 months after enrolment to determine outcomes. The three imaging strategies will be compared regarding subsequent use of healthcare resources over a year. In most large cardiac centres, different imaging modalities are performed by different specialists and therefore an operating grant from one imaging specialty rarely covers the costs of other imaging specialties in comparative studies. To ensure a fair comparison between modalities, all modalities have to be equal. Previous comparative trials have been criticized for being biased towards the technique being promoted by the principal investigator. This trial is unique in that the directors of nuclear cardiology, coronary computed tomography and echocardiography are all specialists in their field and are running state-of-the-art services and were all involved in the early planning of this trial and their involvement has ensured trial design meets clinical need. The results of this trial will give insight into planning of a larger multicentre, multi-national study.

ELIGIBILITY:
Inclusion Criteria:

* Adult Age ≥ 18 years
* Presenting with symptoms suggestive of CAD requiring diagnostic/prognostic workup
* Suitable for Contrast Stress Echocardiography, SPECT and CCTA
* Able and willing to provide consent

Exclusion Criteria:

* Patients with documented CAD (previous invasive angiography, previous STEMI, previous PCI or CABG)
* NSTEMI, ACS within 3 months
* Previous diagnostic imaging tests in the past 6 months
* Women who are pregnant as evidenced by positive pregnancy test
* Breast feeding females
* Significant valvular heart disease (i.e. severe aortic stenosis or regurgitation or severe mitral regurgitation)
* Hemodynamic instability (blood pressure >210/110 ml/Hg or <90/60 mm/Hg)
* Unavailability for follow-up
* Renal insufficiency, eGFR < 30 ml/minute unless on dialysis
* Known allergy to x-ray or echo contrast agents
* Weight exceeding specifications of nuclear equipment (>250 Kg)
* Unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Men and women without known CAD who present with symptoms suggestive of CAD and require diagnostic/prognostic workup.
Sampling Method: Probability Sample
Enrollment: 173 (Actual)
Dates: Start 2012-07; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
healthcare resource utilization | 12 month

SECONDARY OUTCOMES:
referral rates to coronary angiography following three different initial imaging tests in this patient population. | 12 month
coronary lesions which warrant revascularization (including those where it was warranted but not technically possible). | 12 month
radiation exposure from the initial and subsequent imaging procedures | 12 month
total mortality | 12 month
freedom from angina | 12 month
non-fatal myocardial infarction | 12 month
hospital admissions for angina | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: Harald Becher, MD,PhD,FRCP, Principal Investigator — University of Alberta, Alberta Health Services
Locations (1):
- Mazankowski Alberta Heart Institute, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No